CLINICAL TRIAL: NCT03677440
Title: Exercise Training Effects on Cognition and Brain Function in Multiple Sclerosis: A Systematically-Developed Randomized Controlled Trial
Brief Title: Exercise Training Effects on Cognition and Brain Function in Multiple Sclerosis: Project EXACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Brian Sandroff, Principal Investigator, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-300000111; 1R01HD091155-01A1 (NIH)
Record Dates: First submitted 2018-09-14; First posted 2018-09-19 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Cognitive Impairment
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be unaware if the treadmill walking exercise training or stretching-and-toning conditions represent the experimental or control conditions; outcome assessors will be treatment-blinded; MRI data analysts will be blinded to condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill Walking Exercise Training (Experimental): This condition will include 3-months of supervised, progressive light, moderate, and vigorous intensity treadmill walking exercise training based on ACSM guidelines for maximizing adaptations with exercise training. Exercise intensities will be prescribed based on percent oxygen consumption reserve (% VO2R) using values derived from the baseline graded exercise test.
  The exercise training itself will be led by trained exercise leaders who are not involved in the collection of outcome assessments. At the outset of each session, participants will be fitted with a Polar HR Monitor (Oy, Finland), and HR will be monitored continuously throughout each session. Each session will begin with a 5-10 min warm-up, followed by the exercise; the target heart rate reserve (HRR) range associated with the VO2R range will be maintained for as long as possible during each exercise period. This will be followed by a 5-10 min cool-down.
  Interventions: Behavioral: Treadmill Walking Exercise Training
- Stretching-and-Toning Exercise Training (Active Comparator): The active, non-aerobic exercise condition will involve stretching-and-toning activities using the same frequency and duration of the treadmill walking exercise condition. These activities will be based on a manual provided by the National Multiple Sclerosis Society and sessions will be led by trained exercise leaders who are not involved in the collection of outcome assessments. Activities will target the head/neck, shoulder, elbow/forearm, hand/wrist, trunk/hip, ankle/foot. The progression of activities over the 3-month period will involve performing additional exercises and sets along with using progressively thicker elastic resistance bands that provide minimal resistance. Each session is designed to last up to 60 minutes in total. Each session will begin with a warm-up of up to 10 minutes, followed by stretching-and-toning (following the same duration as the treadmill walking exercise training condition) activities, and a cool-down of up to 10 minutes.
  Interventions: Behavioral: Stretching-and-Toning Exercise Training

INTERVENTIONS:
Behavioral: Treadmill Walking Exercise Training — 12-weeks of supervised, progressive treadmill walking exercise training
  Arms: Treadmill Walking Exercise Training
Behavioral: Stretching-and-Toning Exercise Training — 12-weeks of supervised, progressive stretching-and-toning exercise training
  Arms: Stretching-and-Toning Exercise Training

SUMMARY:
Cognitive impairment is highly prevalent, poorly-managed, and disabling in persons with MS and exercise training might represent a promising approach to manage this symptom of the disease. The proposed study aims to examine the effects of 3-months of supervised, progressive (both intensity and duration) treadmill walking exercise training (designed based on pilot work and American College of Sports Medicine guidelines) compared with an active control condition (i.e., stretching-and-toning activities) on cognitive processing speed and functional MRI outcomes in 88 cognitively-impaired persons with MS. This study is critical for providing evidence supporting treadmill walking exercise training as a behavioral approach for managing slowed cognitive processing speed (i.e., the most common MS-related cognitive impairment) and improving brain health in persons with MS.

ELIGIBILITY:
All participants will:

* Be between the ages of 18-65
* Have a clinically definite MS diagnosis based on established criteria
* Be fully-ambulatory based on Expanded Disability Status Scale (EDSS) scores between 0-4.0
* Demonstrate slowed CPS based on initial SDMT scores at least 1 SD below the regression-based normative score for healthy controls (i.e., 16th percentile)
* Be relapse-free and will not have acutely taken corticosteroids for at least 30 days (i.e., relative neurologic stability)
* Not have a history of major depressive disorder, schizophrenia, bipolar disorder I or II, or substance-abuse disorders.
* Not be taking medications that can affect cognition (e.g., antipsychotics, benzodiazepines).
* Be right-handed
* Have corrected vision better than 20/80
* Not have known/diagnosed cardiovascular, metabolic, or renal disease. Individuals with known/diagnosed cardiovascular, metabolic, or renal disease who are asymptomatic will be included only with a physician's approval.
* Demonstrate scores on the Mini-Mental State Examination (MMSE) of 21 or higher (no decisional impairment)
* Be on a stable disease-modifying therapy regimen (i.e., at least 6 months prior to study enrollment).
* Have a low risk for contraindications for MRI based on not having metal (e.g., non-MRI compatible aneurysm clips, metal shards in the body or eyes, or recently placed surgical hardware) or electronic devices (e.g., pacemaker, cochlear implant) within the body.
* Not be pregnant
* Not be engaging in ≥ 150 min of moderate-to-vigorous physical activity (i.e., not meeting public health guidelines for physical activity) per week
* Not be actively engaging in cognitive rehabilitation, or participating in regular brain fitness activities
* Demonstrate systolic blood pressure values of < 200 mmHg or diastolic blood pressure values < 110 mmHg at rest

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Sandroff, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: N=4 participants who were enrolled into the study subsequently dropped out prior to random assignment. Thus, 43 participants were enrolled into the study and 39 participants were randomly assigned into the study arms.
Groups:
- Treadmill Walking Exercise Training: This condition will include 3-months of supervised, progressive light, moderate, and vigorous intensity treadmill walking exercise training based on ACSM guidelines for maximizing adaptations with exercise training. Exercise intensities will be prescribed based on percent oxygen consumption reserve (% VO2R) using values derived from the baseline graded exercise test.
  The exercise training itself will be led by trained exercise leaders who are not involved in the collection of outcome assessments. At the outset of each session, participants will be fitted with a Polar HR Monitor (Oy, Finland), and HR will be monitored continuously throughout each session. Each session will begin with a 5-10 min warm-up, followed by the exercise; the target heart rate reserve (HRR) range associated with the VO2R range will be maintained for as long as possible during each exercise period. This will be followed by a 5-10 min cool-down.
  Treadmill Walking Exercise Training: 12-weeks of supervised, progressive treadmill walking exercise training
Period: Overall Study
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Started | 19 | 20
Completed | 13 | 15
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Population: 2 participants who were enrolled into the study dropped out prior to completing baseline measures
Groups:
- Total: Total of all reporting groups
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.5 (8.0) | 46.1 (11.2) | 45.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 12 | 9 | 21
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 19 | 37
Education [Mean (Standard Deviation); unit: Years] | 16.1 (2.5) | 15.2 (2.2) | 15.6 (2.4)
Expanded Disability Status Scale [Median (Full Range); unit: units on a scale] — This is an ordinal scale of MS disability ranging from 0 (i.e., no disability) to 10 (i.e., death due to MS) that is administered by a Neurostatus-certified examiner. Higher scores indicate worse MS disability.
  units on a scale | 3.0 [2.0 to 4.0] | 3.5 [2.0 to 4.0] | 3.5 [2.0 to 4.0]
Disease Duration [Mean (Standard Deviation); unit: years] | 13.9 (9.9) | 10.9 (7.4) | 11.8 (8.5)
MS Phenotype [Count of Participants; unit: Participants]
  Relapsing-Remitting | 18 | 14 | 32
  Progressive | 0 | 3 | 3
  Unknown | 0 | 2 | 2
Symbol Digit Modalities Test z-score [Mean (Standard Deviation); unit: z-score] — This baseline measure provides an index of MS-related cognitive processing speed impairment using regression-based normative data that accounts for age, sex, and education. A z-score of 0 indicates no impairment relative to healthy controls, accounting for age, sex, and education. Lower z-scores indicate worse MS-related cognitive processing speed impairment.
  z-score | -2.0 (0.7) | -1.9 (0.6) | -1.9 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Processing Speed
Description: Raw (Total) Score from the Symbol Digit Modalities Test (0-110; higher scores indicate faster cognitive processing speed)
Time Frame: Baseline, Follow-up (up to 14 weeks)
Measure: Mean (Standard Deviation); unit: Raw Score
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Number analyzed (Participants) | 13 | 15
Raw Score
  Baseline | 43.5 (9.6) | 43.7 (9.2)
  Follow-up | 46.5 (12.1) | 49.1 (10.7)
Statistical Analysis 1: Comparison: Treadmill Walking Exercise Training vs Stretching-and-Toning Exercise Training; This involves a repeated-measures ANOVA testing a condition (i.e., treadmill walking exercise training vs. stretching-and-toning exercise training)-by-time (i.e., baseline, follow-up) interaction on Symbol Digit Modalities Test scores; Test type: Superiority; p = .34, ANOVA

2. Primary Outcome: Thalamocortical Resting-State Functional Connectivity Region 1
Description: Change in functional connectivity between the thalamus and left superior medial gyrus based on fMRI. As this outcome measure reflects changes in resting-state functional connectivity, positive z-scores indicate increased connectivity and negative z-scores indicate decreased connectivity. A z-score of 0 reflects no change in resting-state functional connectivity.
Time Frame: Follow-up at 12-weeks minus baseline
Population: N=3 participants did not complete MRI at follow-up (12-weeks)
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Number analyzed (Participants) | 11 | 14
z-score | .0334 (.0531) | -.0247 (.0605)
Statistical Analysis 1: Comparison: Treadmill Walking Exercise Training vs Stretching-and-Toning Exercise Training; Test type: Superiority; p = .01, t-test, 1 sided

3. Primary Outcome: Change in Thalamocortical Resting State Functional Connectivity Region 2
Description: Resting-state functional connectivity between the thalamus and left putamen based on fMRI. As this outcome measure reflects changes in resting-state functional connectivity, positive z-scores indicate increased connectivity and negative z-scores indicate decreased connectivity. A z-score of 0 reflects no change in resting-state functional connectivity.
Time Frame: Follow-up at 12-weeks minus baseline
Population: N=3 participants did not complete MRI at follow-up (12-weeks)
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Number analyzed (Participants) | 11 | 14
z-score | .0193 (.0595) | -.0414 (.0783)
Statistical Analysis 1: Comparison: Treadmill Walking Exercise Training vs Stretching-and-Toning Exercise Training; Test type: Superiority; p = .02, t-test, 1 sided

4. Secondary Outcome: 3-second Paced Auditory Serial Addition Test (PASAT)
Description: The 3-second PASAT is a neuropsychological test of working memory, attention, and cognitive processing speed. The total score is the total number of correct answers provided by the participant. The minimum score is 0 and the maximum score is 60. Higher scores reflect better cognition
Time Frame: Baseline, Follow-up (up to 14-weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Number analyzed (Participants) | 12 | 14
score on a scale
  Baseline | 33.8 (16) | 34 (13.4)
  Follow-up | 35.9 (17.0) | 37.4 (13.7)
Statistical Analysis 1: Comparison: Treadmill Walking Exercise Training vs Stretching-and-Toning Exercise Training; Test type: Superiority; p = .63, ANOVA

5. Secondary Outcome: 2-second Paced Auditory Serial Addition Test (PASAT)
Description: The 2-second PASAT is a neuropsychological test of working memory, attention, and cognitive processing speed. The raw score is the total number of correct answers provided by the participant. The minimum score is 0 and the maximum score is 60. Higher scores reflect better cognition.
Time Frame: Baseline, Follow-up (up to 14-weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Number analyzed (Participants) | 12 | 14
score on a scale
  Baseline | 24.8 (13.2) | 25.6 (10.5)
  Follow-up | 26.3 (14.2) | 24.0 (11.5)
Statistical Analysis 1: Comparison: Treadmill Walking Exercise Training vs Stretching-and-Toning Exercise Training; Test type: Superiority; p = .20, ANOVA; Partial eta-squared = .067

6. Secondary Outcome: Pattern Comparison Test
Description: The Pattern Comparison Test is a neuropsychological test of cognitive processing speed wherein participants are asked to specify whether or not two patterns are the same or different. The primary outcome is the total number of correct answers provided by the participant across two 20-second trials. The minimum score is 0 and the maximum score is 60. Higher scores reflect better cognitive processing speed.
Time Frame: Baseline, Follow-up (up to 14-weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Number analyzed (Participants) | 13 | 15
score on a scale
  Baseline | 19.4 (5.6) | 22.1 (5.2)
  Follow-up | 21.3 (5.1) | 24.1 (5.2)
Statistical Analysis 1: Comparison: Treadmill Walking Exercise Training vs Stretching-and-Toning Exercise Training; Test type: Superiority; p = .96, ANOVA

7. Secondary Outcome: Community Integration Questionnaire
Description: The Community Integration Questionnaire is a patient-reported measure of community participation. The minimum score is 0 and the maximum score is 31, with higher scores reflecting better community participation.
Time Frame: Baseline, Follow-up (up to 14-weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline | 19.8 (3.8) | 19.5 (4.2)
  Follow-up | 21.5 (3.6) | 20.5 (3.9)
Statistical Analysis 1: Comparison: Treadmill Walking Exercise Training vs Stretching-and-Toning Exercise Training; Test type: Superiority; p = .55, ANOVA

8. Secondary Outcome: Lawton-Brody Instrumental Activities of Daily Living
Description: The Lawton-Brody Instrumental Activities of Daily Living is a patient-reported measure of the ability to perform instrumental activities of daily living. The minimum score is 0 and the maximum score is 8, with higher scores reflecting a better ability to complete instrumental activities of daily living.
Time Frame: Baseline, Follow-up (up to 14-weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline | 7.7 (0.9) | 7.9 (0.3)
  Follow-up | 8.0 (0.0) | 7.8 (0.4)
Statistical Analysis 1: Comparison: Treadmill Walking Exercise Training vs Stretching-and-Toning Exercise Training; Test type: Superiority; p = .14, ANOVA; Partial eta-squared = .087

9. Secondary Outcome: Multiple Sclerosis Impact Scale-29 Physical Subscale
Description: The Multiple Sclerosis Impact Scale-29 is a patient-reported measure of the impact of multiple sclerosis on physical and mental domains. In this outcome measure, the physical subscale is the component of interest. The minimum score is 0 and the maximum score is 100, with higher scores reflecting greater impact of MS on physical outcomes.
Time Frame: Baseline, Follow-up (up to 14-weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline | 17.9 (16.8) | 23.8 (19.8)
  Follow-up | 11.6 (9.5) | 19.5 (18.9)
Statistical Analysis 1: Comparison: Treadmill Walking Exercise Training vs Stretching-and-Toning Exercise Training; Test type: Superiority; p = .69, ANOVA

10. Secondary Outcome: Timed 25-foot Walk
Description: The timed 25-foot walk is a neuroperformance outcome where participants are asked to walk as quickly and as safely as possible over a 25-foot course free of debris. The primary outcome is the time to walk 25 feet - averaged across two trials. Higher scores reflect slower walking speed and lower scores reflect faster walking speed.
Time Frame: Baseline, Follow-up (up to 14-weeks)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
Number analyzed (Participants) | 12 | 14
Seconds
  Baseline | 5.1 (1.5) | 5.0 (1.0)
  Follow-up | 4.8 (1.1) | 5.1 (1.1)
Statistical Analysis 1: Comparison: Treadmill Walking Exercise Training vs Stretching-and-Toning Exercise Training; Test type: Superiority; p = .28, ANOVA; Partial eta-squared = .048

ADVERSE EVENTS:
Time Frame: 12-weeks
Description: The number of participants at risk for adverse events reflects those who were randomly assigned into the conditions (i.e., n=39).
Arm/Group | Treadmill Walking Exercise Training | Stretching-and-Toning Exercise Training
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 8/19 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treadmill Walking Exercise Training (N=19) | Stretching-and-Toning Exercise Training (N=20)
Minor injury (General disorders) | 5 (5) | 0 (0) — 5 participants experienced minor injuries due to falls that occurred outside of the intervention
Temporary illness (General disorders) | 1 (2) | 1 (1)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Minor Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03677440/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03677440/ICF_001.pdf